CLINICAL TRIAL: NCT00431535
Title: Descriptive Study Concerning the Connection Between SvO2 and Orthostatic Function Post Operatively
Brief Title: Study Concerning Relationship Between Mixed Venous Saturation (SvO2) and Balance
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: SvO2
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2007-10

CONDITIONS: Surgery
Keywords: Fluid; SvO2; Mobilisation; Orthostatic function

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
It is the purpose of the investigators to investigate the possible relationship between fall in the amount of Oxygen in the blood and disturbances of balance-function before and after surgery.

DETAILED DESCRIPTION:
It has been shown that the mixed venous saturation (SvO2) is usable as a parameter of fluid status. It has also been suggested that there is a connection between SvO2 and blood flow in tissue , and that a SvO2 of less than 40% is a sign of tissue hypoxia.

Recently it has been shown that patients going through heart surgery experience a drop in SvO2 during early mobilization.This drop lasts throughout the mobilisation process.

We want to investigate whether the same mechanism applies to patients going through other types of surgery, and whether there is a connection between a drop in SvO2 and orthostatic function.

This will be done by making 3 tests. One pre-operatively,one six hours post-operatively and one 18-24 hours after surgery.

The tests will consist of:

1. 10 min of rest.
2. 3 min of sitting upright on the side of the bed. C. 3 min of standing on the floor. D. 10 min of rest.

Between each position a venous blood sample will be taken. Also 1 blood sample will be taken at the end of surgery.

Continuous measurements by the Finapres system wil be made throughout the test-sequence to investigate changes in BP, SV, TPR and HR.

At the same time the patient will be pain-scored when taking a new position.

ELIGIBILITY:
Inclusion Criteria:

* Patients going through Radical Prostatectomy, where CVC is standard.

Exclusion Criteria:

* Non informed consent
* ASA > II
* Age less than 18, or more than 80 years
* Diabetes Mellitus
* Epidural analgetics
* Alcohol abuse (investigators assessment)
* Unable to understand written or spoken information
* Using beta-blockers

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Joergensen, M.S., Principal Investigator
Locations (2):
- Denmark (2):
  - Dept of anesthesia 2041, ABD centre, Rigshospitalet, Blegdamsvej, Copenhagen, Region Sjælland
  - Rigshospitalet, Copenhagen, Region Sjælland